CLINICAL TRIAL: NCT07376057
Title: Development and Prospective Validation of a Pathology-Based Artificial Intelligence Model for Predicting the Time to Castration Resistance of Prostate Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2025-940-01
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: artificial intelligence; time to castration-resistant; prostate cancer; whole slide image
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Prostatic Neoplasms | interventions — Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Histopathological slides of formalin-fixed, paraffin-embedded tissues from patients with prostate cancer undergoing prostate biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergo prostate biopsy: Patients undergo prostate biopsy and are diagnosed with prostate cancer, who receive Hormone therapy.
  Interventions: Other: Artificial intelligence (AI)-based predictive model (developed)

INTERVENTIONS:
Other: Artificial intelligence (AI)-based predictive model (developed) — Collect pathological slides of prostate biopsy of the enrolled patients. Digitise these slides into whole-slide images (WSIs). Analyze the WSIs using the AI model to generate predictive results (within 12 months, between 12 to 24months or over 24 months). No intervention to patients would be performed in this predictive test study.

SUMMARY:
The goal of this predictive test is to prospectively test the performance of pre-developed artificial intelligence (AI) predictive model for predicting the time to castration resistance of prostate cancer. Investigators had developed this AI model based on deep learning algorithms in preliminary research, and it performed well in retrospective tests.

DETAILED DESCRIPTION:
Hormone therapy is an important treatment method for prostate cancer and can effectively extend the survival of patients. However, almost all patients will progress to castration-resistant prostate cancer at different times. Current Hormone therapy options include androgen deprivation therapy(ADT), anti-androgen receptor(AR), and chemotherapy, with combination therapy being more effective in the early stages but associated with greater side effects. Therefore, predicting the time to castration-resistant progression and using this information to apply personalized treatment plans can ensure efficacy while reducing drug side effects. Therefore, we have developed an artificial intelligence predictive model for predicting the time to castration resistance of prostate cancer, which is expected to accurately predict the progression time for different patients and assist doctors in making personalized and precise treatment plans based on individual progression risks.

This study is a predictive test with no intervention measures, planning to collect pathological slides of prostate biopsy from the enrolled patients and digitise them into whole-slide images (WSIs). The AI model will analyse the WSIs and generate slide-level predictive results (within 12 months, between 12 to 24months or over 24 months). The routine therapy and examination will be performed as usual. These two processes will not interfere with each other. Then we will follow-up the patients for 24 months, to record the time to castration-resistant progression, then we will compare the results with predictive model.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are diagnosed with intermediate- to high-risk prostate cancer; undergo prostate biopsy
2. Patients only received endocrine therapy for prostate cancer;
3. Patients with complete clinical and pathological information.
4. Patients agree to participate in this diagnostic test.

Exclusion Criteria:

1. Patients with other tumors and undergo systemic therapy .
2. The patient refused to participate in this diagnostic test.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prostate cancer, undergo prostate biopsy between Jan, 2026 and Dec 2026 in Sun Yat-sen Memorial Hospital of Sun Yat-sen University are planned to be enrolled in this prospective predictive test. Histopathological slides of biopsy tissues of enrolled patients will be collected and digitised as whole-slide images (WSIs) for prospective validation of the AI model.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
C-index (Concordance Index) | For each enrolled patient, the predictive results of AI model will be obtained in not long after prostate biopsy, and the C-index of the AI model will be evaluated through study completion, an average of 3 year.
  The proportion of all patient pairs in which the predicted outcome order matches the actual outcome order. It estimates the probability that the predicted results are consistent with the observed outcomes.

SECONDARY OUTCOMES:
sensitivity | For each enrolled patient, the predictive results of AI model will be obtained in not long after prostate biopsy, and the sensitivity of the AI model will be evaluated through study completion, an average of 3 year.
  The output of the predictive model is divided into a binary variable using a 12-month threshold: TTCR <12 months is considered a positive outcome, and TTCR ≥12 months is considered a negative outcome. Accordingly, patients with TTCR <12 months are positive patients, and those with TTCR ≥12 months are negative patients. The number of correctly predicted positive slides (TTCR<12 months), to be divided by the number of positive slides in total
specificity | For each enrolled patient, the predictive results of AI model will be obtained in not long after prostate biopsy, and the specificity of the AI model will be evaluated through study completion, an average of 3 year.
  The output of the predictive model is divided into a binary variable using a 12-month threshold: TTCR <12 months is considered a positive outcome, and TTCR ≥12 months is considered a negative outcome. Accordingly, patients with TTCR <12 months are positive patients, and those with TTCR ≥12 months are negative patients. The number of correctly predicted negative slides (TTCR≥12 months), to be divided by the number of negative slides in total

CONTACTS AND LOCATIONS:
Overall Officials: Shaoxu Wu, Ph.D, Study Director — Department of Urology of Sun Yat-sen Memorial Hospital of Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
To protect patient privacy, pathological slide images and other patient-related data are not publicly accessible.